CLINICAL TRIAL: NCT00948597
Title: A Non-Interventional Study to Develop a Pharmacokinetic - Pharmacodynamic Model for Individualized Propofol Dosing
Brief Title: Development of PK/PD Model for Individualized Propofol Dosing
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0721
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Obesity; Elective Surgery
Keywords: propofol; elective surgical procedure; Obese subjects
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participation involves the collection of one blood sample (3.0 ml) in an EDTA (lavender top) tube for pharmacogenetic testing. Genomic DNA will be extracted using standard procedures. Participation in pharmacogenetic testing is optional and requires additional consent; subjects who refuse pharmacogenetifc testing may still be enrolled in this study.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The U.S. National Health and Nutrition Examination Survey of 1994 indicated that 59% of American men and 49% of women have body mass indexes (BMIs) over 25. Extreme obesity, defined as a BMI of 40 or more, was found in 2% of the men and 4% of the women [http://www.cdc.gov/nchs/nhanes.htm]. The newest survey in 2007 indicates an alarming increase in BMI; 63% of Americans are overweight, with 26% now in the obese category. With extreme obesity as high as 26-30% in adults, obesity percentages in children are also sharply on the rise. These alarming numbers pose a major clinical problem in terms of the safe and effective use of drugs in children.

Obesity may alter the disposition and/or clearance of drugs in the body as well as the response, which should be considered when using anesthetics in these patients. Total intravenous anesthesia (TIVA) with propofol is widely used in children, adolescents and adults undergoing surgery, because of rapid onset of action, ease of titration and rapid offset of action. While extensive research on optimal propofol dosing has been performed in non-obese adults, including in critically ill mechanically ventilated adult patients by the investigators' collaborators, there is no evidence on required dosages in morbidly obese adult or pediatric patients of this highly lipophilic agent. As a consequence, serious problems do arise due to under- and overdosing, increasing the risk of inadequate effects and adverse events, respectively. Crucial additional information is needed on the pharmacokinetics of drugs used in morbidly obese children to improve safety and efficacy.

This proposal will test a novel approach by identifying pharmacokinetic/pharmacodynamic (PK/PD) factors that are associated with response to therapy and adverse events. If successful, this study will provide proof of concept data for PK/PD model-based dosing strategy that can be implemented into daily clinical care to allow tailoring of dose to individual needs. Propofol is a versatile anesthetic agent which if dosed to individual needs based on a patient's characteristics and specific PK/PD parameters, will allow individualized dosing, thereby greatly reducing related toxicities. The prospective identification of predictive factors in these morbidly obese high-risk patients represents a new approach to an increasingly common clinical problem. The investigators expect that this study will generate the PK/PD data necessary to continue with a well powered prospective clinical trial.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Hypothesis: The inter-patient variability in propofol effects in relation to clinical response and adverse events in morbidly obese adolescents is associated with identifiable pharmacokinetic factors.

Specific Aim 1: Determine to what extent body weight affects propofol pharmacokinetics (PK) and pharmacodynamics (PD) in morbidly obese adolescents.

Specific Aim 2: Develop a PK/PD model-based dosing algorithm for individualized propofol dosing in morbidly obese adolescents.

To address this hypothesis, we will conduct a clinical study evaluating the pharmacokinetics and pharmacodynamics of propofol in 20 morbidly obese subjects scheduled to undergo laparoscopic gastric banding or another elective procedure. Full PK/PD profiles will be obtained during surgery and the Bispectral index monitor will be used as a validated approach for PD monitoring, a measure of depth of anesthesia (5). The population nonlinear mixed effect modeling (NONMEM) approach will be used with extensive covariate analysis to account for observed inter- and intraindividual variability (6, 7). The potential covariates affecting propofol PK (and PD) we will explore include total body weight, lean body mass, Body Mass Index (BMI), Body Surface Area (BSA), height, age, gender, type of procedure, and duration of procedure.

In addition, in an exploratory fashion, we will evaluate propofol pharmacogenetics. CYP2B6 and UGT1A9 are highly polymorphic enzyme responsible for the metabolism of propofol (20, 21). Novel allelic forms of CYP2B6 (22) and UGT1A9 (23) were identified recently that potentially could explain some of the large between patient variability in clearance resulting in large differences in propofol blood concentrations and responses to standard doses.

STUDY DESIGN Description of Study Design The study will be a clinical non-intervention study and will not interfere with the standard anesthetic and perioperative care except for BIS monitoring and additional blood sampling from an indwelling line during and following anesthesia. One blood sample for genetic testing (3 ml) and 1.0 ml for baseline PK/PD modeling will be drawn from a venous line placed for clinical standard of care. The remaining 1.0 ml serial blood samples for pharmacokinetic modeling will be drawn from an indwelling venous line placed under anesthesia.

The rate that propofol will be given will be standardized to minimize variability between anesthesiologists. Induction of anesthesia will be done with an infusion of 1000mcg/kg/min of propofol. This bolus will be followed by propofol infusion at a rate of 250-350 mcg/kg/min for 10 min, and then titrated to clinical needs by the anesthesia team.

Propofol Concentration Measurements: Blood samples (1.0 ml) will be collected from an indwelling line in oxalate tubes. Samples will be collected at scheduled time points. The number of samples for subjects may vary depending on the amount of time subjects are in surgery. Samples may also be drawn at unscheduled time points if propofol dose adjustments are made during the surgical procedure. The total sample volume for propofol concentration measurements will not exceed 22ml.

Samples will be collected at the following scheduled and unscheduled time-points. Times for sample collection are approximations. Ideally, samples beginning with the 15 minute collection should be obtained within +/- 5 minutes of the times listed, when possible:

Scheduled time points:

Baseline:

• within 15 minutes prior to induction of propofol

After induction of propofol:

* 1-3 min
* 5 min
* 10 min

  * 15 min
  * 30 min
  * 45 min
  * 60 min
  * 120 min
  * 180 min
  * 240 min
  * Within 5 min prior to stopping propofol infusion

After the end of propofol infusion

* 5 min
* 10 min
* 15 min
* 30 min
* 45 min
* 120 min

Unscheduled time points:

* Within 5 min prior to each dose adjustment
* 60 min after each dose adjustment

NOTE: If a scheduled sample collection falls within 10 minutes of an unscheduled sample collection, only the unscheduled sample will be collected.

Whole blood samples will be stored at 4°C until analysis (within 1 month).

BIS Monitoring: An age and head size-appropriate disposable BIS sensor (standard pediatric or XP sensor, Aspect Medical Systems, Norwood, MA) will be placed on each child's forehead and will be connected to a BIS monitor as directed by the manufacturer and described recently by us (5). The sensors are single-use and are latex/PVC free.

Each sensor contains a strip of electrodes. This one-piece unit is coated with a medical grade adhesive to establish electrical contact when placed on the forehead, and is designed for symmetrical placement to capture bi-hemispheric data. The sensor is attached via a cable to a VISTA stand alone unit module that serves as an interface between the sensor and the BIS monitor. This module is a signal converter, which acquires the electroencephalogram (EEG) signal from the sensors and converts the EEG signal to digital format. The EEG signal is then processed and the BIS index is played on the monitor. Data output (processed and raw EEG) will be downloaded.

The BIS monitor screen will be covered during the procedure to ensure that anesthesia personnel involved in the care will be blinded to the BIS score and trend screen to avoid BIS score influenced changes in propofol doses. At the end of the procedure, the BIS data will be electronically transferred to a computer along with time points and other study parameters (18). Data that will be collected on case report forms include the following: date and time of BIS data collection, including start and end times; minimum, average and maximum BIS values at various time points including during propofol bolus doses, rate changes and discontinuation; average Signal Quality Index (SQI);and average electromyography (EMG).

Demographic and Clinical Data: We will use and analyze patient demographic and clinical data in combination with the PK/PD data (10, 11) for Pharmacokinetic /Pharmacodynamic modeling purposes. Patient data to be collected include: age, gender, ethnicity, weight, height and body mass index. Clinical data to be collected and recorded on case report forms include: blood pressure, heart rate, temperature and end tidal carbon dioxide level (ETCO2). Other clinical data that will be recorded on case report forms include: time needed to lose consciousness (loss of verbal contact), start/stop time of propofol dosing, propofol infusion rates, propofol dose adjustments, time to eye opening on verbal command post infusion, and sedation scores (Ramsey sedation scale) post-operatively every 10 minutes (+/- 2 minutes) for the first 30 minutes and thereafter every 30 minutes (+/- 5 minutes) while in the Post Anesthesia Care Unit (PACU).

Pharmacogenetics: Participation involves the collection of one blood sample (3.0 ml) in an EDTA (lavender top) tube for pharmacogenetic testing. Genomic DNA will be extracted using standard procedures.

Questionnaire(s): The Structured Awareness Screening Interview shall be used to detect awareness during the anesthetic period which can be an adverse event related to underdosing/reduced sensitivity to propofol effects (24). This questionnaire has been used to detect awareness and perioperative behavioral studies for children age 5 and older (25). The same questions will be used for all children. No incentives will be given for the children to answer, and no leading questions will be asked during the screening interview.

For this study, the questionnaire will be administered two times, on post-operative day (POD) 1 and 3. The POD1 questionnaire will be administered by a study anesthesiologist. If the subject answers "no" on question six, the anesthesiologist may decide to not continue the interview. For subjects discharged prior to POD 3, parents or a legal representative will be given a written set of questions before leaving the hospital and will be requested to ask their child the questions on POD 3, write down the child's responses, and mail the questions back. To justify repeated questioning, the parents will be told that a child's memories of their anesthetic might change with time. They shall be instructed to ask the questions exactly as they are written and to write down their child's reply verbatim. If a child answers the POD3 questions directly instead of being asked the questions by a parent, their responses will be evaluated for inclusion by the Principal Investigator. Subjects consented as adults may answer the questions directly.

If a subject is still in the hospital on POD 3, a study anesthesiologist will administer the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 5 to 18 years of age;
* Have a Body Mass Index (BMI) greater than 30;
* Be scheduled for bariatric or other elective surgical procedure;
* Will be administered propofol anesthesia as part of procedure and standard of care and subject is expected to be under anesthesia for at least 60 minutes;
* Signed and dated IRB-approved Informed Consent or Parental Permission and Assent form, as applicable.

Exclusion Criteria:

* Patients receiving investigational agent as part of another clinical study;
* Patients with severe developmental delay, known neurological disorders;
* Conditions where the placement of the sensor or process of assessment could interfere with the BIS monitoring;
* Allergy to propofol / anaphylaxis to egg protein;
* History of severe sleep apnea;
* Anticipated difficult airway access;
* Significant allergies and sensitivities to tape and/or adhesives.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from the Cincinnati Children's Hospital Medical Center Surgical Weight Loss Program for Teens (Thomas Inge, Director), supplemented with general surgery patients who are overweight and have a Body Mass Index (BMI) of more than 30.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in propofol clearance and volume of distribution (for determination of effective concentration); Depth of anesthesia. | Samples will be analyzed within one month of collection

SECONDARY OUTCOMES:
Population PK/PD model (NON-MEM) using patient demographic and clinical data. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A Vinks, PharmD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Diepstraten J, Chidambaran V, Sadhasivam S, Esslinger HR, Cox SL, Inge TH, Knibbe CA, Vinks AA. Propofol Clearance in Morbidly Obese Children and Adolescents : Influence of Age and Body Size. Clin Pharmacokinet. 2012 Aug;51(8):543-551. doi: 10.1007/BF03261930. PMID 28258392
- [Derived] Chidambaran V, Venkatasubramanian R, Sadhasivam S, Esslinger H, Cox S, Diepstraten J, Fukuda T, Inge T, Knibbe CAJ, Vinks AA. Population pharmacokinetic-pharmacodynamic modeling and dosing simulation of propofol maintenance anesthesia in severely obese adolescents. Paediatr Anaesth. 2015 Sep;25(9):911-923. doi: 10.1111/pan.12684. Epub 2015 May 13. PMID 25975390
- [Derived] Diepstraten J, Chidambaran V, Sadhasivam S, Esslinger HR, Cox SL, Inge TH, Knibbe CA, Vinks AA. Propofol clearance in morbidly obese children and adolescents: influence of age and body size. Clin Pharmacokinet. 2012 Aug 1;51(8):543-51. doi: 10.2165/11632940-000000000-00000. PMID 22690673